CLINICAL TRIAL: NCT06538649
Title: Determining the Therapeutic Potential of Statins on Stricturing Crohn's Disease
Brief Title: Effect of Statins on Crohn's Disease
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Sidhartha Ranjit Sinha, Assistant Professor of Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 76686
Record Dates: First submitted 2024-08-01; First posted 2024-08-06 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2024-12

CONDITIONS: Crohn's Ileocolitis; Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Intervention Model Description: Random assignment (2:1) to either statin (Arm 1) or placebo (Arm 2), such that 2/3 of participants will be assigned to Arm 1, and 1/3 of participants will be assigned to Arm 2.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Statin (Experimental): Rosuvastatin tablet(s) once daily for 6-12 months. Dose will start at 10 mg daily (5 mg daily for Asians), then increase to 20 mg for those tolerating and without contraindication.
  Interventions: Drug: Rosuvastatin
- Control (Placebo Comparator): Placebo tablet(s) taken once daily for 6-12 months.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Rosuvastatin — Rosuvastatin provided at 10 mg start; 5mg for Asians. Dose will be increased to 20 mg for those tolerating and without contraindication.
  Other Names: Crestor
  Arms: Statin
Other: Placebo — Placebo tablet(s)
  Arms: Control

SUMMARY:
The goal of this clinical trial is to learn if statins work to prevent strictures in adults with Crohn's disease. The main question it aims to answer is:

* Can statins reduce the formation of strictures in participants with stricturing Crohn's disease?

Researchers will compare statins to a placebo (a look-a-like substance that contains no drug) to see if statins work to prevent strictures from forming. Participants will:

* Take statins or a placebo every day for 6-12 months
* Visit the clinic for lab tests twice after starting either statins or placebo
* Complete questionnaires about symptoms and medications
* Respond to monthly check-ins (via phone call) during participation

DETAILED DESCRIPTION:
Strictures are a formidable complication of Crohn's disease (CD), with more than half of patients experiencing clinically significant bowel obstructions. Stricturing CD is a primary driver of morbidity and hospital admissions and is frequently associated with treatment failures. Moreover, it is estimated that nearly 50% of patients with CD will undergo bowel resection surgery within ten years of diagnosis, highlighting the severity and persistence of this issue for patients as well as the healthcare system.

By modulating inflammatory and fibrotic pathways, the investigators posit that statins reduce primary stricture development and also recurrence after stricture resection.

The investigators will assess the impact of statin therapy on early stricture recurrence in a pilot, randomized controlled clinical trial in patients undergoing stricture resection, evaluating both clinical outcomes and detailed immune, microbiome, and metabolic profiling. Through this effort, the investigators will determine if statins reduce clinical and biological signs of stricture recurrence in the short term.

ELIGIBILITY:
Inclusion Criteria:

1. Established diagnosis of stricturing Crohn's disease
2. Scheduled for surgical resection of terminal ileum strictures at either

   * Stanford University, or
   * Dr. Phillip Fleshner's colorectal surgery practice in Los Angeles

Exclusion Criteria:

1. Pregnant, nursing, or planning to become pregnant in the next 6-12 months
2. Severe renal dysfunction (stage 5 chronic kidney disease (CKD), end-stage renal disease (ESRD))
3. Known clinical allergy or prior adverse reaction to statin therapy (e.g., rhabdomyolysis)
4. Current use of cyclosporine
5. Current use of statin therapy prior to study initiation
6. Clinical diagnosis of active liver disease (beyond metabolic dysfunction-associated steatotic liver disease (MASLD)) with unexplained persistent elevations in hepatic transaminase levels
7. Current use of any of the following medications, without explicit clearance from a treating physician to enroll in the study:

   * Antifungals (e.g., ketoconazole, itraconazole, voriconazole)
   * Fibrate drugs
   * Macrolide antibiotics (e.g., erythromycin, clarithromycin)
   * Protease inhibitors (e.g., ritonavir, lopinavir)
   * Calcium channel blockers (e.g., verapamil, diltiazem)
   * Amiodarone
   * Warfarin
   * Colchicine

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Rutgeerts score | 6-12 months post surgery
  Will be assessed at post surgery surveillance colonoscopy. Minimum score is i0 (no lesions) and maximum score is i4 (diffuse inflammation with already larger ulcers, nodules and/or narrowing), with higher scores meaning a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Sidhartha R Sinha, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No